CLINICAL TRIAL: NCT03586089
Title: PHENObarbital for the MANagement of Severe Acute ALcohol Withdrawal Syndrome (PHENOMANAL): a Prospective Randomized Feasibility Study.
Brief Title: Phenobarbital for Severe Acute Alcohol Withdrawal Syndrome
Acronym: PHENOMANAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting patients
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-285
Record Dates: First submitted 2018-06-21; First posted 2018-07-13 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Alcohol Withdrawal Delirium; Alcohol Withdrawal; Alcohol Withdrawal Seizures
Keywords: Phenobarbital; Alcohol; Withdrawal
MeSH Terms: conditions — Alcohol Withdrawal Delirium; Alcohol Withdrawal Seizures | interventions — Phenobarbital; Diazepam

STUDY DESIGN:
Intervention Model Description: As soon as possible after randomization, patients will receive either a single IV dose of phenobarbital (7.5 mg per kg of ideal body weight, prepared in 250 ml D5W; n=26) or placebo (250 ml D5W; n=13)
Who Masked: Participant, Care Provider, Investigator
Masking Description: To conceal allocation, central randomization will be conducted by the Pharmacy Department of Unity Health Toronto - St. Michael's Hospital using a list of random treatment assignments created on www.randomize.net.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phenobarbital (Experimental): Patients will receive a single dose of phenobarbital (7.5 mg/kg of ideal body weight, IV) in addition to usual therapy.
  Interventions: Drug: Phenobarbital Sodium
- Placebo (Placebo Comparator): Patients will receive an inactive placebo (IV).
  Interventions: Drug: Inactive placebo

INTERVENTIONS:
Drug: Phenobarbital Sodium — Single IV dose of phenobarbital (7.5 mg per kg of body weight prepared in 250 ml D5W)
  Other Names: Symptom-triggered benzodiazepines (e.g., Valium)
  Arms: Phenobarbital
Drug: Inactive placebo — Single dose of inactive placebo prepared in 250 ml D5W).
  Other Names: Symptom triggered benzodiazepines (e.g., Valium)
  Arms: Placebo

SUMMARY:
Severe acute alcohol withdrawal syndrome is a potentially life-threatening condition characterized by agitation, confusion, abnormal heart rhythms and seizures. Typically, clinicians treat the symptoms of alcohol withdrawal with a class of medications known as benzodiazepines (e.g., Valium). These medications have a short duration of activity and require repeated administration, often every hour or less, to reduce the symptoms of alcohol withdrawal. Many patients suffer complications related to inadequate treatment of alcohol withdrawal (e.g., abnormal heart rhythms, aspiration, seizures) resulting in admission to an intensive care unit and prolonged hospital stay, all of which increase healthcare costs. Although alcohol withdrawal is common, especially among disadvantaged (e.g., homeless) patients, limited funding is available to advance the care of patients suffering from alcohol withdrawal. A safe and effective treatment for severe alcohol withdrawal would benefit patients and our healthcare system.

Phenobarbital is an inexpensive, commonly available medication that is typically used to treat seizures. A key advantage of phenobarbital is that its calming effect lasts for a long period of time and it can be given as a 'one-time-dose' intravenously, so that it both prevents and treats withdrawal symptoms and reduces the need for repeated benzodiazepines. Through better symptom control, phenobarbital is expected to reduce the costs and complications of alcohol withdrawal. At present, physicians rarely use phenobarbital for this purpose, and additional research is needed for this medication to become part of routine care in clinical practice.

The PHENOMANAL pilot trial will assess safety and whether clinicians can administer a single dose of phenobarbital intravenously, in addition to benzodiazepines, compared to benzodiazepines alone for treating patients with severe alcohol withdrawal. This information will inform the design of a larger clinical trial. For patients, the PHENOMANAL trial has the potential to revolutionize how patients suffering from severe alcohol withdrawal are treated. For society and the healthcare system, phenobarbital is expected to reduce the complications and costs associated with severe alcohol withdrawal.

DETAILED DESCRIPTION:
In a 39 patient, single-centre pilot trial of phenobarbital as an adjunctive treatment for severe acute alcohol withdrawal syndrome (AAWS), the PHENOMANAL trial will demonstrate the ability to recruit, consent, and randomize participants and adhere to the assigned treatment protocol with minimal loss to follow up and infrequent adverse events. This pilot trial will provide data and proof of feasibility in preparation to conduct a multicentre randomized controlled trial of phenobarbital as an adjunctive treatment for severe AAWS. Patients will be recruited from the Emergency Department, Intensive Care Unit, Medical Step-Up unit, and wards of Unity Health Toronto - St. Michael's Hospital, a quaternary care centre located in downtown Toronto, Canada.

Recruitment Patients will be identified by research personnel during daytime hours from Monday to Friday using a multi-modal approach. With the assistance of the hospital informatics department, personnel will collect a daily census of patients who have been started on symptom-triggered benzodiazepine therapy using the Clinical Institute Withdrawal Assessment (revised) (CIWA-Ar) protocol.

Consent The investigators will use a hybrid consent model. Whenever possible, consent will be obtained from the patient or his/her substitute-decision-maker (SDM) at the time of recruitment. In this instance, Research Coordinators will ask one of the members within the 'circle of care' (e.g., physician, nurse, respiratory technologist, social worker, etc) to ask for permission from patient or their SDM for a research coordinator to contact him/her about participation in research.

Randomization To conceal allocation, central randomization will be conducted by the Pharmacy Department of St. Michael's Hospital using a list of random treatment assignments created on www.randomize.net.

Intervention As soon as possible after randomization, patients will receive either a single intravenous (IV) dose of phenobarbital (7.5 mg per kg of ideal body weight, prepared in 250 ml D5W; n=26) or placebo (250 ml D5W; n=13).

Safety During the infusion patients will be monitored with continuous oximetry, non-invasive blood pressure measurement q 30 minutes (+/-, and continuous cardiac monitoring in a high-acuity unit (e.g Intensive Care, Cardiac Intensive Care, Emergency, Step-Up). Phenobarbital achieves peak serum concentration within one hour of administration; however, study participants will be monitored with continuous pulse oximetry and q 30 minute non-invasive blood pressure measurement for a minimum of 3 hours post administration. Each patient will thus receive a total of four hours of intensive monitoring (i.e. one hour of monitoring during the study drug administration, and three hours of monitoring subsequently to ensure clinical stability). Eligible female trial participants < 55 years of age will have a urine or blood ßhCG checked prior to treatment administration.

Data Collection Research personnel will collect data on (i) Patient Demographics including age; sex; housing; relevant comorbidities; time since last alcohol consumption; baseline laboratory investigations; and baseline CIWA-Ar scores. (ii) Treatment including maximal CIWA-Ar score; number, dose and type of benzodiazepine or alternative treatments administrated (e.g., benzodiazepines, propofol, clonidine, dexmedetomidine, haloperidol); vital signs; need for admission to a monitored setting (i.e. vitals recorded more often than every 4 hours, or need for continuous oximetry); use of non-invasive or invasive ventilation; and the presence of a bedside sitter. These data will be recorded for a span of 7 days or until hospital discharge (whichever comes first). (iii) Clinical Outcomes including adverse events (aspiration, intubation, seizures); monitored care and hospital length of stay; time to Addictions Medicine assessment; and vital status at hospital discharge.

Statistical Power Fifty patients will be recruited in the PHENOMANAL pilot trial. This sample size will ensure that clinicians gain experience with the treatment protocol, enable assessment of recruitment and consent practices, and provide preliminary estimates of treatment effect (safety and efficacy) to inform the design of a larger trial.

Statistical Analysis In the primary analysis, recruitment will be considered feasible if the investigators can recruit 2 or more patients per month, on average, over the 24-month study period. In secondary analyses, compliance rates greater than 80% will be considered acceptable in both study arms. Similarly, a cross-over rate of < 10% from the control arm to the phenobarbital arm will be taken to be acceptable. Preliminary estimates of treatment effect will be compared between the alternative treatment strategies using the Chi-Squared test (alternatively, Fisher's Exact test) and Student's T-test (Alternatively, Wilcoxon Rank-Sum test) for binary and continuous data, respectively.

Discussion This pilot randomized controlled trial will assess feasibility of a multicenter trial to investigate intravenous phenobarbital as an adjunctive treatment for severe AAWS. Randomization of 39 patients will allow us to assess feasibility metrics, including clinicians' ability to comply with the protocol and cross-over rates, and generate preliminary estimates of safety and treatment effect.

This trial protocol has been designed in light of the unique challenges of studying patients with severe AAWS. It is important to clearly define the population of interest. Patients with mild alcohol withdrawal may not benefit from IV adjunctive treatment with phenobarbital, and may lead to over-sedation, complications (e.g., intubation, aspiration), and/or prolonged hospitalization. Oral phenobarbital administration may warrant further investigation in this patient population. In contrast, highly agitated patients suffering from AAWS may not show a clinically important response to the dose of IV phenobarbital that the investigators are evaluating. The investigators decision to limit enrollment to patients with a severely elevated CIWA score (>16) after receiving at least 60 mg of diazepam or equivalent represents an attempt identify the patient population that is most likely to benefit from treatment with adjunctive IV phenobarbital. Base on pharmacokinetics, phenobarbital is most likely to be useful if administered early in the course of treatment and thus enrollment will be accordingly limited to the first 16 hours after patients are identified.

ELIGIBILITY:
Inclusion Criteria:

1. Alcohol withdrawal syndrome (regardless of admitting diagnosis).
2. Severe symptoms, as defined by a 'Clinical Institute for Withdrawal Assessment Adult revised' (CIWA-Ar) score of 16 or more, or delirium severe enough to prohibit assessment with the CIWA-Ar, or observed withdrawal seizures, in each case despite treatment with at least 60 mg of diazepam (or an equivalent dose of another benzodiazepine) in the previous 16 hours, regardless of route of administration..
3. Early alcohol withdrawal, broadly defined as the first 16 hours after the diagnosis of acute alcohol withdrawal has been made. The time of diagnosis will be taken to be the time of prescription of symptom-triggered benzodiazepine therapy ("CIWA protocol"), or the time of consultation to ICU/Emergency Department, Internal Medicine, or the Addictions Service (Psychiatry) for the management of alcohol withdrawal.
4. Anticipated need for hospitalization (i.e. admission to ICU, medical step-up unit, or wards).

Exclusion Criteria:

1. an alternate etiology for delirium thought to be more likely than alcohol withdrawal;
2. age <16 years;
3. pregnancy (positive assay for ßhCG). A urine assay or blood test will be performed for all women < 55 yrs;
4. current breastfeeding;
5. severe acute hepatitis (AST or ALT >500); liver failure (INR >2 not otherwise explained);
6. a presenting complaint of neurotrauma, brain mass, or intra-cranial bleed; abnormal cell count or gram stain on lumbar puncture (if performed);
7. strong clinical suspicion of recent co-ingestion of depressant drugs (e.g. opioids, toxic alcohols, gamma-hydroxy-butyrate);
8. hemodynamic instability (systolic blood pressure [SBP] < 90 mmHg);
9. history of barbiturate allergy;
10. history of porphyria;
11. history of myasthenia gravis;
12. inability to obtain IV access;
13. anticipated transfer to another centre;
14. stated intent to leave against medical advice;
15. active outpatient prescription for anti-retroviral therapy for HIV
16. active outpatient prescription for one of the following anti-epileptic drugs: valproic acid, phenytoin, carbamazepine, clobazam, lacosamide, lamotrigine, levetiracetam, topiramate, primidone, or phenobarbital.
17. active outpatient prescription for an anticoagulant medication with a significant metabolic interaction with phenobarbital (i.e. warfarin or apixaban).
18. active outpatient prescription for a monoamine oxidase inhibitor (e.g., phenelzine, selegiline, tranylcypromine, isocarboxazid)
19. renal failure, as defined by a creatinine clearance <10 mls/minute (as calculated by Cockcroft-Gault equation) and/or active receipt of renal replacement therapy (dialysis).
20. administration of IV or oral phenobarbital during the index admission prior to randomization.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Safety: adverse event rate | 18 months
  The rates of severe adverse events, including aspiration events and endotracheal intubation, will be compared between treatment and placebo groups.

SECONDARY OUTCOMES:
Protocol feasibility: recruitment rate | 18 months
  In the primary analysis, we will consider recruitment feasible if we can recruit 2 to 3 patients per month, on average, over the 18-month study period.

OTHER OUTCOMES:
Protocol adherence: crossover rate | 18 months
  In secondary analyses, we will consider compliance rates greater than 80% to be acceptable in both study arms. Similarly, we will consider a cross-over rate of < 10% from the control arm to the phenobarbital arm to be acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Burns, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Filewod N, Hwang S, Turner CJ, Rizvi L, Gray S, Klaiman M, Buell D, Ailon J, Caudarella A, Ginocchio GF, Santos M, Sandhu G, Dewhurst N, Sequeira K, Burns KEA. Phenobarbital for the management of severe acute alcohol withdrawal (the PHENOMANAL trial): a pilot randomized controlled trial. Pilot Feasibility Stud. 2022 Jan 22;8(1):14. doi: 10.1186/s40814-021-00963-4. PMID 35065662